CLINICAL TRIAL: NCT05587452
Title: Early Screening of Colorectal Cancer Based on Plasma Multi-omics Combining With Artificial Intelligence-a Multi-center, Prospective Study
Brief Title: Early Screening of Colorectal Cancer Based on Plasma Multi-omics Combining With Artificial Intelligence
Acronym: RECOMMEND
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: Cangzhou Central Hospital (Other); Weifang Medical University (Other); Heji Hospital affiliated to Changzhi Medical College (Unknown); Beijng Fengtai Hospital (Unknown)
Responsible Party: Principal Investigator, Jianqiang Tang, Associate professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Other Study IDs: NCC3511
Record Dates: First submitted 2022-10-17; First posted 2022-10-20 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Colorectal Adenoma; Colorectal Cancer
Keywords: Colorectal cancer; Early screening; Multi-omics; ctDNA; Artifical intelligence
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy group: People without colorectal adenoma or cancer
  Interventions: Diagnostic Test: Colonoscopy; Diagnostic Test: Test of ctDNA methylation; Diagnostic Test: Test of characteristics of ctDNA fragment
- Advanced adenoma group: People with colorectal adenoma
  Interventions: Diagnostic Test: Colonoscopy; Diagnostic Test: Test of ctDNA methylation; Diagnostic Test: Test of characteristics of ctDNA fragment
- Colorectal cancer group: People with colorectal cancer
  Interventions: Diagnostic Test: Colonoscopy; Diagnostic Test: Test of ctDNA methylation; Diagnostic Test: Test of characteristics of ctDNA fragment

INTERVENTIONS:
Diagnostic Test: Colonoscopy — Colonoscopy is performed to identify whether the patient has colorectal adenoma or cancer
Diagnostic Test: Test of ctDNA methylation — A specified panel is used to detect the site of methylation of ctDNA in plasma
Diagnostic Test: Test of characteristics of ctDNA fragment — Low pass whole genome sequencing is used to detect the characteristics of ctDNA fragment

SUMMARY:
To evaluate the accuracy and effectiveness of a novel screening method based on plasma multi-omics combining with artificial intelligence in a large prospective cohort for the detection of colorectal cancer and advanced adenomas.

DETAILED DESCRIPTION:
Minimally invasive detection of circulating tumor DNA (ctDNA) in peripheral blood of patients with colorectal malignancies via liquid biopsy has emerged as a promising biomarker. This is urgently needed, as conventional imaging and plasma protein-derived biomarkers lack sensitivity and specificity.The goal of this observational study is to evaluate the effectiveness and accuracy of a novel screening method based on plasma multi-omics combining with artificial intelligence in five hospitals around China for the detection of colorectal cancer and advanced adenomas.

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion criteria for colorectal cancer/advanced adenoma 1) Voluntarily participate and sign the informed consent form, and be able to cooperate with the entire research process 2) Be able to provide sufficient and qualified blood samples for this study 3) Patients with pathological diagnosis of colorectal cancer stage I-III (TNM staging according to AJCC 8th edition colorectal cancer staging system) 4) No previous cancer treatment, including chemotherapy, radiotherapy, targeted or immunotherapy, and any surgery treat 5) Advanced adenoma should at least meet one of the following conditions: ① Diameter >10mm ② Villus-tubiform adenoma ③ More than 25% of villi structure in mixed adenoma ④High-grade intraepithelial neoplasia
2. Inclusion criteria for healthy people 1) Voluntarily participate and sign the informed consent form, and be able to cooperate with the entire research process 2) Diagnosed without colorectal adenoma or cancer by colonoscopy within 12 months

Exclusion Criteria:

1. Exclusion criteria for colorectal cancer/advanced adenoma 1) Women who are pregnant or breastfeeding 2) Currently diagnosed with another cancer or have a history cancer 3) Persistent fever or receiving anti-inflammatory treatment within 14 days before blood samples are taken in this study 4) Receiving blood transfusion within 30 days 5) Receiving organ transplantation or previous non-autologous (allogeneic) bone marrow or stem cell transplantation 6) Digestive tract bleeding, obstruction, perforation and any trauma or surgery within 3 months 7) Poor physical condition, not suitable for extraction blood samples 8) Subjects who are judged by the investigator to be unsuitable to participate in this study for other reasons;
2. Exclusion criteria for healthy people 1) Women who are pregnant or breastfeeding 2) Receiving organ transplantation or previous non-autologous (allogeneic) bone marrow or stem cell transplantation 3) Have a history cancer 4) Receiving blood transfusion within 30 days 5) Poor physical condition, not suitable for extraction Blood samples 6) Diagnosed with precancerous lesions by colonoscopy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Heathy group: Patients without colorectal adenoma or cancer examined by colonoscopy Precancerous group: Patients at least meet one of the following conditions: ① Diameter >10mm ② Villus-tubiform adenoma ③ More than 25% of villi structure in mixed adenoma ④High-grade intraepithelial neoplasia Colorectal cancer group: Patients diagnosed with adenocarcinoma by colonoscopy and histological examination.
Sampling Method: Non-Probability Sample
Enrollment: 950 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | Through study completion, an average of 1 year
  Sensitivity (for colorectal cancer and\or advanced precancerous neoplasm) of this plasm-based multi-omics test. The diagnostic colonoscopy procedure is reference method. Lesions will be confirmed as malignancy or precancerous by pathological biopsy.
Specificity | Through study completion, an average of 1 year
  Specificity (for colorectal cancer and\or advanced precancerous neoplasm) of this plasm-based multi-omics test. The diagnostic colonoscopy procedure is reference method. Lesions will be confirmed as malignancy or precancerous by pathological biopsy.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beiijing Fengtai Hospital, Beijing, Beijing Municipality
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - Affiliated Hospital of Weifang Medical University, Weifang, Shandong
  - Heji Hospital affiliated to Changzhi Medical College, Changzhi, Shanxi